CLINICAL TRIAL: NCT00420953
Title: A Randomized, Double-blind, 2-period Crossover Trial to Determine the Relative Bioavailability of PM101 I.V. (Amiodarone HCl) and Cordarone I.V. in Healthy Adult Volunteers
Brief Title: Relative Bioavailability of PM101 IV and Cordarone IV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prism Pharmaceuticals (Industry)
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Healthy
MeSH Terms: interventions — Amiodarone

INTERVENTIONS:
Drug: Cordarone

SUMMARY:
Determine the relative bioavailability of PM101 I.V. and Cordarone I.V.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male or female 18 to 59 years of age, inclusive. Women of childbearing potential must be using a medically acceptable form of birth control for the duration of the trial and must have a negative serum pregnancy test at screening and upon check-in to the study facility.
* Have a BMI within the range of 18-35 kg/m2, inclusive.
* Be able to communicate effectively with the study personnel.
* Have no significant disease or abnormal laboratory values as determined by medical history, physical examination or laboratory evaluations, conducted at the screening visit or on admission to the clinic.
* Have a normal 12-lead electrocardiogram, without any clinically significant abnormalities of rate, rhythm or conduction and including normal QTc segment time, i.e. <430 for males and <450 for females.
* Be nonsmokers defined as not having smoked in the past 6 months prior to dosing.
* Be adequately informed of the nature and risks of the study and give written informed consent prior to receiving study medication.

Exclusion Criteria:

* Known hypersensitivity or allergy to Cordarone I.V. or its excipients.
* Known hypersensitivity or allergy to iodine or radio-opaque dyes.
* Women who are pregnant or breast feeding.
* A history or presence of asthma or other pulmonary disease, thyroid disease (hypo- or hyperthyroidism), hepatitis or other liver disease.
* Any disease or condition (medical or surgical) which, in the opinion of the investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk.
* The presence of abnormal laboratory values which are considered clinically significant.
* Positive screen for Hepatitis B (HbsAg, Hepatitis B Surface Antigen), Hepatitis C (anti HCV, Hepatitis C Antibody), or HIV (anti-HIV 1/2).
* Received an investigational drug within a period of 30 days prior to enrollment in the study.
* Received any drug therapy within 2 weeks prior to administration of the first dose of any study-related treatment. This exclusion is extended to 4 weeks for any drugs known to induce or inhibit hepatic drug metabolism.
* Consumption of alcohol within 48 hours prior to dose administration or during any in-patient period.
* A positive urine drug screen including ethanol, cocaine, THC, barbiturates, amphetamines, benzodiazepines, and opiates.
* Any history of alcohol abuse, illicit drug use (use of soft drugs [such as marijuana] within 3 months prior to screening visit or hard drugs [such as cocaine, phencyclidine [PCP] and crack] within 1 year prior to the screening visit), significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction.
* A history of difficulty with donating blood.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows: 50 mL to 499 mL of whole blood within 30 days, or more than 499 mL of whole blood within 56 days prior to drug administration.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-12-18 (Actual); Primary Completion 2007-04-23 (Actual); Study Completion 2007-04-23 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability and safety

CONTACTS AND LOCATIONS:
Locations (1):
- Anapharm, Montreal, Quebec, Canada